CLINICAL TRIAL: NCT06698757
Title: Eight Vs Four Cycles of Preoperative Neoadjuvant Sintilimab in Mismatch-repair Deficient/microsatellite Instability-high, Locally Advanced Colorectal Cancer(OPEN): a Multi-center, Open-label, Prospective Randomized Controlled Trial
Brief Title: Different Cycles of Preoperative Neoadjuvant Sintilimab in Mismatch-repair Deficient/microsatellite Instability-high, Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yugui Lian (Other)
Responsible Party: Sponsor-Investigator, Yugui Lian, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-1330-003
Record Dates: First submitted 2024-11-09; First posted 2024-11-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8 cycles of neoadjuvant treatment with Sintilimab (Experimental): A total of 48 subjects were enrolled and received Sintilimab at a dose of 200 mg, administered via intravenous infusion on the first day of each cycle, with each cycle lasting 3 weeks (Q3W), for a total of 8 treatment cycles.
  Interventions: Biological: Sintilimab
- 4 cycles of neoadjuvant treatment with Sintilimab (Active Comparator): A total of 48 subjects were enrolled and received Sintilimab at a dose of 200 mg, administered via intravenous infusion on the first day of each cycle, with each cycle lasting 3 weeks (Q3W), for a total of 4 treatment cycles.
  Interventions: Biological: Sintilimab

INTERVENTIONS:
Biological: Sintilimab — Subjects were enrolled and received Sintilimab at a dose of 200 mg, administered via intravenous infusion on the first day of each cycle, with each cycle lasting 3 weeks (Q3W)

SUMMARY:
Colorectal cancer is one of the most common malignant tumors, accounting for approximately 10% of new cancer cases and cancer-related deaths worldwide each year. In recent years, with the development of industrialization and urbanization, the increase in the number of elderly patients, and changes in dietary structure and lifestyle habits, the incidence and mortality rates of colorectal cancer in China have risen significantly. Some patients are already in locally advanced or late stages at the time of diagnosis, making treatment more difficult. Among them, patients with MSI-H/dMMR colorectal cancer account for about 10% to 15% of the total.

Neoadjuvant therapy for rectal cancer primarily targets resectable mid-to-low rectal cancer patients with T3/4 and any N stage. Currently, neoadjuvant therapy for rectal cancer mainly involves chemoradiotherapy, while patients with a low risk of recurrence may opt for neoadjuvant chemotherapy. For patients with mid-to-low locally advanced rectal cancer, intensified systemic chemotherapy can be chosen before and after preoperative radiotherapy. For patients with technical difficulties in sphincter preservation but a strong desire to preserve the sphincter, higher intensity treatments can be considered, such as the CinClare protocol of concurrent chemoradiotherapy with capecitabine and irinotecan, the FOWARC protocol of concurrent radiotherapy with FOLFOX, or interval chemotherapy, including total neoadjuvant therapy. However, for MSI-H/dMMR patients, neoadjuvant chemoradiotherapy is less effective. Xu Ruihua from the Sun Yat-sen University Cancer Center evaluated the clinical response and safety of four cycles of neoadjuvant treatment with sintilimab in dMMR or MSI-H colorectal cancer. In this study, 16 patients underwent at least one response evaluation. All six patients who underwent radical surgery achieved R0 resection. Tumor shrinkage was observed in 15 patients (94%) at the first evaluation after treatment. Among the 16 evaluable patients, 3 (19%) underwent radical surgery and achieved pCR, 9 (56%) achieved cCR and opted for a watch-and-wait strategy, 3 (19%) did not achieve cCR and underwent radical surgery with residual tumor found in the pathological specimens. One patient (6%) discontinued treatment due to a severe adverse event (grade 3 encephalitis), did not achieve cCR, and refused surgery. The results of immunotherapy in patients with MSI-H/dMMR metastatic colorectal cancer have greatly encouraged researchers to explore its application in neoadjuvant therapy. The NICHE study, the world's first neoadjuvant immunotherapy study in non-metastatic colon cancer, showed a 100% MPR and a 69% pCR rate after neoadjuvant immunotherapy in 32 patients with dMMR colon cancer. Based on this study, the larger NICHE-2 study was conducted, enrolling a total of 112 patients with non-metastatic dMMR colon cancer. These patients received one dose of ipilimumab (1 mg/kg) combined with nivolumab (3 mg/kg) followed by one dose of nivolumab (3 mg/kg) monotherapy within 6 weeks before surgery. The short-term efficacy results showed an MPR of 95% and a pCR rate of 67%, consistent with previous results, with good tolerability and only 4% experiencing grade 3-4 adverse events.

Sintilimab targets the same molecule as nivolumab and pembrolizumab but has a different amino acid sequence. Multiple preclinical in vitro studies have validated the effect of sintilimab in blocking the PD-1 pathway. Completed preclinical pharmacodynamics, animal pharmacokinetics, and toxicology studies have shown that sintilimab has clear targets, reliable cell line sources, good drug stability, and has demonstrated good activity in completed preclinical studies.

Based on multiple previous studies, the optimal cycle for neoadjuvant immunotherapy has not yet been determined. However, different treatment cycles result in significant differences in pCR, which may be related to the number of treatment cycles. This study aims to explore the postoperative pathological complete response rate of 8 cycles versus 4 cycles of neoadjuvant sintilimab treatment in dMMR/MSI-H locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* has pathologically confirmed colon cancer or upper rectal cancer (with the lower edge of the tumor more than 10 cm from the anal verge); clinical stage cT3/T4 or N+
* no urgent need for surgery due to bleeding, perforation, or obstruction
* immunohistochemistry of tumor biopsy indicating deficient mismatch repair (dMMR), defined by the loss of expression of one or more of the four proteins MSH1, MSH2, MSH6, and PMS2; or genetic testing indicating MSI-H

Exclusion Criteria:

* Has distant metastatic disease.
* Has received prior medical therapy (chemotherapy, immunotherapy, biologic, or targeted therapy), radiation therapy or surgery for management of colon cancer
* Has undergone any major surgical procedure, open biopsy, or experienced significant traumatic injury within 28 days prior to randomization
* Is receiving any other anticancer or experimental therapy. No other experimental therapies (including but not limited to chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, or other experimental drugs) of any kind are permitted while the participant is receiving study intervention
* There is a history of illness or evidence of disease, treatment, or abnormal laboratory test values that could potentially interfere with the trial results or hinder the subject's full participation in the study, or any other conditions deemed unsuitable for inclusion by the investigator.
* The investigator believes there are other potential risks that make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2031-11-15 (Estimated)

PRIMARY OUTCOMES:
the pathological complete response rate (pCR) | From randomization up to a median of 5 years after randomization.
  Evaluate the pathological complete response rate (pCR) after surgery in patients with locally advanced dMMR/MSI-H colorectal cancer who received 4 cycles versus 8 cycles of neoadjuvant treatment with sintilimab.

SECONDARY OUTCOMES:
Event-free Survival (EFS) | From randomization up to a median of 5 years after randomization.
  EFS is defined as the time from randomization to either disease recurrence or death due to any cause or treatment related toxicity that results in the participant not being suitable for surgery
Overall Survival (OS) | From randomization up to a median of 5 years after randomization.
  OS is defined as time from randomization to death from any cause
Number of Participants with treatment emergent adverse events (AEs), serious adverse events (SAEs), Immune-mediated Adverse Event (imAEs), AEs leading to death and AEs leading to discontinuation of study treatment | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zheng'zhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.